CLINICAL TRIAL: NCT00600145
Title: Dose Response of Mirtazapine to Methamphetamine Induced Interest, Mood Elevation and Reward
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision
Sponsor: University of Virginia (Other)
Collaborators: American Association of Chairs of Departments of Psychiatry (Other)
Responsible Party: Gabrielle Marzani-Nissen, MD, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13222
Record Dates: First submitted 2008-01-10; First posted 2008-01-24 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Amphetamine Dependence
Keywords: Human volunteers; amphetamine dependence
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Mirtazapine
  Interventions: Drug: Mirtazapine
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mirtazapine — 15 mg Mirtazapine is administered followed 2 hours later by 20 mg of methamphetamine / placebo (administered at each testing visit)
  Other Names: Remeron
  Arms: 1
Other: Placebo — Placebo
  Arms: 2

SUMMARY:
The primary purpose of this study is to determine if Mirtazapine will produce a decrease in interest in the drug, a decrease in mood elevation, and/or a decrease in reward when given before methamphetamine compared to placebo.

Participants will be screened with a psychiatric interview, medical history and physical, laboratory tests, drug of abuse screen and, if female, a urine pregnancy test. They will be provided written informed consent. They will be studied in a within-subjects examination of the subjective mood responses of mirtazapine and methamphetamine. Interactions between methamphetamine and mirtazapine will be assessed by pharmacokinetic studies. Each participant will be introduced to rating scales and cognitive tasks described below. Participants will remain in the research unit for 5 hours on each day that they receive study medication or placebo. They will spend five days in total on the research unit, one day separated by at least one day; then in two day blocks separated by at least one day from another two day block. A venous catheter will be placed for blood draws. Blood pressures and heart rates will be recorded and assessed. Participants will be randomized and double blinded to receive either placebo or mirtazapine orally two hours prior to the administration of randomized and double blinded methamphetamine or placebo in order to have the peak effects of the drugs overlap. VAS-mood, ARCI, GRS, POMS and POMS-E, neurocognitive tasks Trails A and B and Symbol digits modalities test will be administered prior to the mirtazapine or placebo dose, and repeated after the administration of methamphetamine or placebo. After the administration of methamphetamine or placebo, vital signs will be assessed every 15 minutes and the measures will be repeated until 120 minutes have passed from the initial dose of methamphetamine or placebo. Blood will be drawn at one, three and four hour marks for pharmacokinetic testing. This will be repeated on each testing day.

DETAILED DESCRIPTION:
Methamphetamine dependence is a major health problem in the US. Methamphetamine's reinforcing effects associated with its abuse liability depend upon activation of the cortico-mesolimbic dopamine (CMDA) system. Medications that antagonize CMDA function might have therapeutic potential Mirtazapine appears to affect this pathway. Mirtazapine works through serotinergic (5-HT) mechanisms 5HT 2 and 3, alpha 2 and H1 antagonist and has been noted to decrease excitatory responses in methamphetamine challenged animals. Mirtazapine increases dopamine release in the prefrontal cortex by 5HT receptor activation. Additionally, in a randomized, placebo controlled trial; individuals taking mirtazapine for amphetamine detoxification were found to have significant improvements in hyper arousal and anxiety subset score when discontinuing the stimulant. Methamphetamine has been given safely to healthy human volunteers in other studies.

We propose to conduct the first preliminary human laboratory study to determine if mirtazapine 15 mg diminishes methamphetamine (20 mg) induced positive subjective interest, mood elevation and reinforcing value. This dose of methamphetamine has been used by other investigators in healthy volunteers.

This preliminary trial is the first in a sequence of studies to characterize the dose dependent effects of mirtazapine as a treatment agent for methamphetamine dependence. If this study is successful, it would afford us a scientific platform and rationale for progressing with testing efficacy for mirtazapine among methamphetamine dependent individuals both in the human laboratory and in clinical trials. The primary objective of this study is to evaluate systematically the neurobehavioral basis and dose-response effects of mirtazapine acutely on methamphetamine-induced interest, mood elevation and reward. This study employs a well-validated, state-of-the-art, human laboratory technique to determine the extent to which mirtazapine blocks methamphetamine induced euphoria, reinforcement, and cue craving in healthy volunteers tested in a controlled hospital environment under medical supervision.

ELIGIBILITY:
Inclusion Criteria:

* 18 -45 years old
* healthy human volunteers
* no history of pre-existing physical (including cardiovascular) illness
* no history of drug abuse or dependence (defined below)
* ability to read and write

Exclusion Criteria:

* pregnant
* any psychotropic medication
* criteria for active substance abuse or dependence based on the DSM-IV: For substance abuse: A maladaptive pattern of substance use leading to clinically significant impairment or distress, as manifested by one (or more) of the following, occurring within a 12-month period:

  1. recurrent substance use resulting in a failure to fulfill major role obligations at work, school, home (e.g., repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; neglect of children or household)
  2. recurrent substance use in situations in which it is physically hazardous (e.g., driving an automobile or operating a machine when impaired by substance use)
  3. recurrent substance-related legal problems (e.g., arrests for substance-related disorderly conduct)
  4. continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (e.g., arguments with spouse about consequences of intoxication, physical fights)
* The symptoms have never met the criteria for Substance Dependence for this class of substances.
* For substance dependence: A maladaptive pattern of substance use, leading to clinically significant impairment or distress, as manifested by three (or more) of the following, occurring at any time in the same 12-month period:

  1. tolerance, as defined by either of the following:

     1. a need for markedly increased amounts of the substance to achieve intoxication or desired effect
     2. markedly diminished effect with continued use of the same amount of substance
  2. withdrawal, as manifested by either of the following:

     1. the characteristic withdrawal syndrome for the substance
     2. the same (or a closely related) substance is taken to relieve or avoid withdrawal symptoms
  3. the substance is often taken in larger amounts or over a longer period than was intended
  4. there is a persistent desire or unsuccessful efforts to cut down or control substance use
  5. a great deal of time is spent in activities to obtain the substance, use the substance, or recover from its effects
  6. important social, occupational or recreational activities are given up or reduced because of substance use
  7. the substance use is continued despite knowledge of having a persistent or recurrent physical or psychological problem that is likely to have been caused or exacerbated by the substance (e.g., continued drinking despite recognition that an ulcer was made worse by alcohol consumption) on any stimulant medication including:

     * Amphetamine (Adderall®, Adderall XR®)
     * Dextroamphetamine (Dexedrine®)
     * Methamphetamine (Desoxyn®)
     * Dexmethylphenidate (Focalin®, Focalin® XR)
     * Diethylpropion (Tenuate®, Tenuate Dospan®)
     * Methylphenidate (Metadate CD®, Ritalin LA®, Methylin®, Ritalin®, Metadate ER®, Ritalin SR®, Methylin ER®, Daytrana®, Concerta®)
     * Pemoline (Cylert®)
     * Benzphetamine (Didrex®)
     * Phendimetrazine (Adipost®, Bontril®, Melfiat®, Prelu-2®, X-Trozine LA®, Bontril PDM®, Obezine®, Obezine caplets) ®
     * Phentermine (Ionamin®, Phentride®, Teramine®, Adipex-P®)
     * Sibutramine (Meridia®)
     * Caffeine (No Doz®, Quick-Pep®, Vivarin®, Caffedrine®,Caffeine and sodium benzoate inj, Cafcit®)
     * Doxapram (Dopram®)
     * Modafinil (Provigil®)
     * Cocaine
     * MDMA (Ecstasy)
     * MDA
* history of hypertension (BP > 140/90 mm Hg) or systolic hypotension (BP <90/75 mm Hg).
* Subjects with resting pulse rate >90/min.
* any active medical illness
* Subjects known to have clinically significant medical conditions, as determined by complete physical examination, or, a past or current history of the following conditions (including but not limited to):
* cerebrovascular accident or transient ischemic attack;
* ischemic heart disease or myocardial infarction;
* symptomatic coronary artery disease or peripheral vascular disease;
* malignancy or history of malignancy within the past 5 years (except basal cell carcinoma);
* renal disease and/or impaired renal function as defined by subjects with a creatinine clearance of £60 ml/min/24hrs;
* diseases of the gastrointestinal system including active liver disease or current active hepatitis;
* subjects with AST and/or ALT >2 times the upper limit of the normal range and/or an increased serum bilirubin >2 times the upper limit of normal at screening;
* pulmonary disorders
* endocrinological disorders including thyroid disorders;
* gross neurological disorders including subjects with seizure disorders and subjects with progressive or degenerative neurological disorders (e.g., multiple sclerosis)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
extent to which mirtazapine reduces methamphetamine induced mood elevation, reward, and interest | At each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle Marzani-Nissen, MD, Principal Investigator — University of Virginia
Locations (1):
- Universiyt of Virginia, Charlottesville, Virginia, United States